CLINICAL TRIAL: NCT05786859
Title: The Efficacy and Safety of Rifaximin In The Treatment of HBV Associated Acute-on-Chronic Liver Failure Patients With Mild to Moderate Hepatic Encephalopathy
Brief Title: The Efficacy and Safety of Rifaximin Treatment
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, The Efficacy and Safety of Rifaximin In The Treatment of HBV Associated Acute-on-Chronic Liver Failure Patients With Mild to Moderate Hepatic Encephalopathy., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Efficacy of Rifaximin
Record Dates: First submitted 2023-03-12; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Liver Failure, Acute on Chronic; Hepatic Encephalopathy; HBV; Hepatitis B; Rifaximin; Effect of Drug
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatic Encephalopathy; Hepatitis B | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Single center randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin Treatment Group (Experimental)
  Interventions: Drug: Rifaximin 200 mg
- Standard Treatment Group (control group) (Sham Comparator)
  Interventions: Other: Standard Treatment without Rifaximin

INTERVENTIONS:
Drug: Rifaximin 200 mg — Rifaximin Treatment Group:on the basis of comprehensive treatment of liver failure, Rifaximin will be added, three times a day, 400mg each time, for a total of 4 weeks, and we will observe until 12 weeks after withdrawal.
  Arms: Rifaximin Treatment Group
Other: Standard Treatment without Rifaximin — The standard treatment group (control group), which will receive routine comprehensive treatment for liver failure without Rifaximin.
  Arms: Standard Treatment Group (control group)

SUMMARY:
There will be 124 patients diagnosed as hepatitis B associated acute on chronic liver failure with mild to moderate hepatic encephalopathy will be enrolled in this study according to the inclusion and exclusion criteria, and will be randomly divided into two groups as 1:1.First group is called Rifaximin group, on the basis of comprehensive treatment of liver failure, Rifaximin (Alfa Sigma S.p.A) is added, three times a day, 400 mg each time, for a total of 4 weeks, and observed until 12 weeks after withdrawal. The other group is called standard treatment group (control group), which will receive routine comprehensive treatment for liver failure. The reversal of mild to moderate hepatic encephalopathy in the two groups of patients will be observed within 4 weeks, then follow up to 12 weeks.

DETAILED DESCRIPTION:
Liver failure is a common clinical syndrome of severe liver disease, with a high mortality rate. On the basis of chronic liver disease, acute on chronic liver failure is a syndrome characterized by acute jaundice deepening and coagulation dysfunction caused by various inducements, which can be combined with hepatic encephalopathy, ascites, electrolyte disorder, infection, hepatorenal syndrome, hepatopulmonary syndrome and other complications, as well as extrahepatic organ failure. At present, the medical treatment of acute on chronic liver failure is still lacks of efficient drugs and means. On the other hand, the mortality rate of liver transplantation can be as high as 50-70%. The occurrence of bacterial infection, hepatic encephalopathy, hepatorenal syndrome and other complications is significantly related to the high mortality of acute on chronic liver failure. Common causes of liver failure include hepatitis virus, drugs or hepatotoxic substances, autoimmune diseases, etc. In China, hepatitis B virus infection is the main cause of acute on chronic liver failure.

Previous studies have confirmed that intestinal flora imbalance and translocation are important reasons for decompensated cirrhosis complicated with primary bacterial peritonitis. Gram-positive bacteria (including enterococcus, staphylococcus, etc.) and multidrug resistant bacteria have become common pathogenic bacteria of spontaneous bacterial peritonitis. A randomized controlled clinical study on spontaneous bacterial peritonitis in Europe shows that gram-positive bacteria account for 62.5% of bacteria isolated from ascites, enterococcus accounted for the majority. The intestinal flora imbalance and translocation are also important inducements of decompensated cirrhosis complicated with hepatic encephalopathy and hepatorenal syndrome. Patients with acute on chronic liver failure also have intestinal flora imbalance. Recent research shows that the proportion of enterococci in hepatitis B associated acute on chronic liver failure is significantly increased, and during the progress of hepatitis B associated acute on chronic liver failure, enterococcus faecium rapidly increases, which is related to poor prognosis. Due to the severe inflammatory reaction, patients with acute on chronic liver failure are prone to intestinal barrier function defects. Therefore, intestinal flora imbalance and translocation are closely related to the complications of acute on chronic liver failure complicated by bacterial infection and hepatic encephalopathy.

Rifaximin- α (referred to as Rifaximin) is a drug that is not easy to be absorbed and only works locally in the gastrointestinal tract. The concentration in the intestinal tract is much higher than MIC90 of the intestinal flora. It has broad-spectrum antibacterial activity, can cover gram-positive and gram-negative bacteria, and is not conducive to the screening of drug-resistant strains. The efficacy and safety of Rifaximin in the prevention and treatment of hepatic encephalopathy in patients with decompensated cirrhosis have been confirmed by many large randomized controlled clinical trials worldwide, and it is the only drug approved by FDA in the United States for the treatment and prevention of hepatic encephalopathy in the past 30 years. Over the past 10 years, experimental and clinical evidence has shown that Rifaximin may have other beneficial effects on the course of liver cirrhosis by regulating intestinal microflora and affecting the gut-liver axis. Rifaximin has been reported for the prevention of other complications of cirrhosis, including spontaneous bacterial peritonitis, hepatorenal syndrome, reduction of portal pressure, prevention of bleeding from esophageal varices, and treatment of refractory ascites in cirrhosis.

In the drug information about Rifaximin released by the FDA of the United States, it was mentioned that patients with severe liver damage (Child-Pugh C) should be cautious in use, because in the clinical experiment of using rifaximin to prevent and treat hepatic encephalopathy, it was found that rifaximin 550 mg/time, twice a day, for patients with Child-Pugh score A, B and C, the amount of drugs entering the systemic circulation was 10 times higher than that of the healthy control group (12.3 ± 4.8 ng • h/mL), 14 times and 21 times (257 ± 100.2 ng • h/mL).Therefore, most previous clinical trials only included patients with MELD score less than 25. Although the systemic exposure of patients with severe liver damage was higher than that of the healthy control group, due to the low total exposure, the side effects of Rifaximin were rare in the clinical study of decompensated cirrhosis, and the incidence of adverse events was similar to that of the control group. Because Rifaximin mainly takes effect locally in the intestine, the systemic bioavailability is low, and the safety data of Rifaximin in patients with liver cirrhosis, FDA does not recommend adjusting the dose for patients with severe liver damage, and the drug instructions also indicate that dose adjustment is not necessary for patients with liver insufficiency.

A recently published multicenter exploratory study suggested that the use of rifaximin in patients with severe alcoholic hepatitis (MELD score 19-24) was safe, and compared with the control group, the use of Rifaximin could reduce the incidence of infection and the incidence of infection-related acute on chronic liver failure after the use of glucocorticoids in severe alcoholic hepatitis. However, the safety and efficacy of Rifaximin in patients with hepatitis B (HBV) associated acute on chronic liver failure have not been reported. Our study plans to evaluate the safety and effectiveness of Rifaximin in the treatment of hepatitis B(HBV) associated acute on chronic liver failure complicated with mild to moderate hepatic encephalopathy through a randomized controlled study.

There will be 124 patients diagnosed as hepatitis B associated acute on chronic liver failure with mild to moderate hepatic encephalopathy will be enrolled in this study according to the inclusion and exclusion criteria, and will be randomly divided into two groups as 1:1.First group is called Rifaximin group, on the basis of comprehensive treatment of liver failure, Rifaximin (Alfa Sigma S.p.A) is added, three times a day, 400 mg each time, for a total of 4 weeks, and observed until 12 weeks after withdrawal. The other group is called standard treatment group (control group), which will receive routine comprehensive treatment for liver failure. The reversal of mild to moderate hepatic encephalopathy in the two groups of patients will be observed and recorded within 4 weeks, then follow up to 12 weeks. The occurrence of various complications related to liver failure and survival situation will be recorded within 12 weeks, during this time, serum of the two groups of patients will be collected, and the changes of biochemical and coagulation indicators and the changes of serum bacterial translocation-related markers will be recorded. The feces of patients before and after treatment will be collected for intestinal microecological analysis.

ELIGIBILITY:
1. Inclusion Criteria:

   * The confirmed HBsAg positive patients with chronic hepatitis B are defined as HBsAg positive for at least 6 months or evidence of chronic HBV infection;
   * Acute onset, progressive deepening of jaundice, serum total bilirubin (TB) ≥ 85umol/L and severe coagulation dysfunction, international standardized ratio (INR) ≥ 1.5 or plasma prothrombin activity (PTA)<40%
   * The score of the psychological test scale of hepatic encephalopathy is less than - 4 points or mild to moderate (degree I or II) manifestations of hepatic encephalopathy, including the decline of computational ability, timing and orientation, personality change, lethargy, and positive flapping wing tremor.
   * Be able and willing to provide informed consent and comply with the test requirements.
2. Exclusion Criteria:

   * There are definite infections or hepatorenal syndromes during screening;
   * Upper gastrointestinal bleeding occurred within 1 week before screening;
   * Have used sedative drugs such as "benzodiazepines" or other psychotropic drugs within one week before screening;
   * Those with severe primary heart, lung, kidney and other important organ dysfunction affecting life expectancy;
   * HIV infection;
   * Uncontrolled malignant tumor, nerve and mental abnormality;
   * Patients who are allergic to the study drugs and excipients;
   * Pregnant or lactating women;
   * In the late stage of liver failure, MELD score>35;
   * Other circumstances in which the researcher believes that the patient should not participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The reversal rate of hepatic encephalopathy between 2 groups in 4 weeks. | 4 weeks
  The reversal rate of hepatic encephalopathy in the 2 groups within 4 weeks will be recorded.

SECONDARY OUTCOMES:
The incidence of complications related to liver failure within 12 weeks between 2 groups. | 12 weeks
  The incidence of complications related to liver failure will be recorded in the 2 groups during 12 weeks.
The survival rate between 2 groups within 12 weeks. | 12 weeks
  The survival rate will be observed in the two groups within 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarin SK, Choudhury A, Sharma MK, Maiwall R, Al Mahtab M, Rahman S, Saigal S, Saraf N, Soin AS, Devarbhavi H, Kim DJ, Dhiman RK, Duseja A, Taneja S, Eapen CE, Goel A, Ning Q, Chen T, Ma K, Duan Z, Yu C, Treeprasertsuk S, Hamid SS, Butt AS, Jafri W, Shukla A, Saraswat V, Tan SS, Sood A, Midha V, Goyal O, Ghazinyan H, Arora A, Hu J, Sahu M, Rao PN, Lee GH, Lim SG, Lesmana LA, Lesmana CR, Shah S, Prasad VGM, Payawal DA, Abbas Z, Dokmeci AK, Sollano JD, Carpio G, Shresta A, Lau GK, Fazal Karim M, Shiha G, Gani R, Kalista KF, Yuen MF, Alam S, Khanna R, Sood V, Lal BB, Pamecha V, Jindal A, Rajan V, Arora V, Yokosuka O, Niriella MA, Li H, Qi X, Tanaka A, Mochida S, Chaudhuri DR, Gane E, Win KM, Chen WT, Rela M, Kapoor D, Rastogi A, Kale P, Rastogi A, Sharma CB, Bajpai M, Singh V, Premkumar M, Maharashi S, Olithselvan A, Philips CA, Srivastava A, Yachha SK, Wani ZA, Thapa BR, Saraya A, Shalimar, Kumar A, Wadhawan M, Gupta S, Madan K, Sakhuja P, Vij V, Sharma BC, Garg H, Garg V, Kalal C, Anand L, Vyas T, Mathur RP, Kumar G, Jain P, Pasupuleti SSR, Chawla YK, Chowdhury A, Alam S, Song DS, Yang JM, Yoon EL; APASL ACLF Research Consortium (AARC) for APASL ACLF working Party.. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific association for the study of the liver (APASL): an update. Hepatol Int. 2019 Jul;13(4):353-390. doi: 10.1007/s12072-019-09946-3. Epub 2019 Jun 6. PMID 31172417
- [Result] Wong F, Piano S, Singh V, Bartoletti M, Maiwall R, Alessandria C, Fernandez J, Soares EC, Kim DJ, Kim SE, Marino M, Vorobioff J, Barea RCR, Merli M, Elkrief L, Vargas V, Krag A, Singh SP, Lesmana LA, Toledo C, Marciano S, Verhelst X, Intagliata N, Rabinowich L, Colombato L, Kim SG, Gerbes A, Durand F, Roblero JP, Bruns T, Yoon EL, Girala M, Pyrsopoulos NT, Kim TH, Yim SY, Juanola A, Gadano A, Angeli P; International Club of Ascites Global Study Group. Clinical features and evolution of bacterial infection-related acute-on-chronic liver failure. J Hepatol. 2021 Feb;74(2):330-339. doi: 10.1016/j.jhep.2020.07.046. Epub 2020 Aug 8. PMID 32781201
- [Result] Wiest R, Lawson M, Geuking M. Pathological bacterial translocation in liver cirrhosis. J Hepatol. 2014 Jan;60(1):197-209. doi: 10.1016/j.jhep.2013.07.044. Epub 2013 Aug 28. No abstract available. PMID 23993913
- [Result] Dever JB, Sheikh MY. Review article: spontaneous bacterial peritonitis--bacteriology, diagnosis, treatment, risk factors and prevention. Aliment Pharmacol Ther. 2015 Jun;41(11):1116-31. doi: 10.1111/apt.13172. Epub 2015 Mar 26. PMID 25819304
- [Result] Piano S, Fasolato S, Salinas F, Romano A, Tonon M, Morando F, Cavallin M, Gola E, Sticca A, Loregian A, Palu G, Zanus G, Senzolo M, Burra P, Cillo U, Angeli P. The empirical antibiotic treatment of nosocomial spontaneous bacterial peritonitis: Results of a randomized, controlled clinical trial. Hepatology. 2016 Apr;63(4):1299-309. doi: 10.1002/hep.27941. Epub 2015 Aug 4. PMID 26084406
- [Result] Bajaj JS, Khoruts A. Microbiota changes and intestinal microbiota transplantation in liver diseases and cirrhosis. J Hepatol. 2020 May;72(5):1003-1027. doi: 10.1016/j.jhep.2020.01.017. Epub 2020 Jan 28. PMID 32004593
- [Result] Wang K, Zhang Z, Mo ZS, Yang XH, Lin BL, Peng L, Xu Y, Lei CY, Zhuang XD, Lu L, Yang RF, Chen T, Gao ZL. Gut microbiota as prognosis markers for patients with HBV-related acute-on-chronic liver failure. Gut Microbes. 2021 Jan-Dec;13(1):1-15. doi: 10.1080/19490976.2021.1921925. PMID 34006193
- [Result] Jiang ZD, Ke S, Palazzini E, Riopel L, Dupont H. In vitro activity and fecal concentration of rifaximin after oral administration. Antimicrob Agents Chemother. 2000 Aug;44(8):2205-6. doi: 10.1128/AAC.44.8.2205-2206.2000. PMID 10898704
- [Result] Bass NM, Mullen KD, Sanyal A, Poordad F, Neff G, Leevy CB, Sigal S, Sheikh MY, Beavers K, Frederick T, Teperman L, Hillebrand D, Huang S, Merchant K, Shaw A, Bortey E, Forbes WP. Rifaximin treatment in hepatic encephalopathy. N Engl J Med. 2010 Mar 25;362(12):1071-81. doi: 10.1056/NEJMoa0907893. PMID 20335583
- [Result] Sidhu SS, Goyal O, Mishra BP, Sood A, Chhina RS, Soni RK. Rifaximin improves psychometric performance and health-related quality of life in patients with minimal hepatic encephalopathy (the RIME Trial). Am J Gastroenterol. 2011 Feb;106(2):307-16. doi: 10.1038/ajg.2010.455. Epub 2010 Dec 14. PMID 21157444
- [Result] Caraceni P, Vargas V, Sola E, Alessandria C, de Wit K, Trebicka J, Angeli P, Mookerjee RP, Durand F, Pose E, Krag A, Bajaj JS, Beuers U, Gines P; Liverhope Consortium. The Use of Rifaximin in Patients With Cirrhosis. Hepatology. 2021 Sep;74(3):1660-1673. doi: 10.1002/hep.31708. Epub 2021 Jun 7. PMID 33421158
- [Result] Elfert A, Abo Ali L, Soliman S, Ibrahim S, Abd-Elsalam S. Randomized-controlled trial of rifaximin versus norfloxacin for secondary prophylaxis of spontaneous bacterial peritonitis. Eur J Gastroenterol Hepatol. 2016 Dec;28(12):1450-1454. doi: 10.1097/MEG.0000000000000724. PMID 27512927
- [Result] Goel A, Rahim U, Nguyen LH, Stave C, Nguyen MH. Systematic review with meta-analysis: rifaximin for the prophylaxis of spontaneous bacterial peritonitis. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1029-1036. doi: 10.1111/apt.14361. Epub 2017 Oct 9. PMID 28994123
- [Result] Ibrahim ES, Alsebaey A, Zaghla H, Moawad Abdelmageed S, Gameel K, Abdelsameea E. Long-term rifaximin therapy as a primary prevention of hepatorenal syndrome. Eur J Gastroenterol Hepatol. 2017 Nov;29(11):1247-1250. doi: 10.1097/MEG.0000000000000967. PMID 28902040
- [Result] Zeng X, Sheng X, Wang PQ, Xin HG, Guo YB, Lin Y, Zhong JW, He CZ, Yin J, Liu TT, Ma WJ, Xiao X, Shi PM, Yuan ZL, Yang L, Ma X, Xu JM, Shen XZ, Yang CQ, Zhu X, Lv NH, Xie WF. Low-dose rifaximin prevents complications and improves survival in patients with decompensated liver cirrhosis. Hepatol Int. 2021 Feb;15(1):155-165. doi: 10.1007/s12072-020-10117-y. Epub 2021 Jan 1. PMID 33385299
- [Result] Lv XY, Ding HG, Zheng JF, Fan CL, Li L. Rifaximin improves survival in cirrhotic patients with refractory ascites: A real-world study. World J Gastroenterol. 2020 Jan 14;26(2):199-218. doi: 10.3748/wjg.v26.i2.199. PMID 31988585
- [Result] Jimenez C, Ventura-Cots M, Sala M, Calafat M, Garcia-Retortillo M, Cirera I, Canete N, Soriano G, Poca M, Simon-Talero M, Altamirano J, Lucey M, Garcia-Tsao G, Brown RS Jr, Schwabe RF, Verna EC, Schnabl B, Bosques-Padilla F, Mathurin P, Caballeria J, Louvet A, Shawcross DL, Abraldes JG, Genesca J, Bataller R, Vargas V. Effect of rifaximin on infections, acute-on-chronic liver failure and mortality in alcoholic hepatitis: A pilot study (RIFA-AH). Liver Int. 2022 May;42(5):1109-1120. doi: 10.1111/liv.15207. Epub 2022 Mar 7. PMID 35220659
- See also: Related Info — https://www.accessdata.fda.gov/drugsatfda_docs/label/2017/021361s023lbl.pdf